CLINICAL TRIAL: NCT05147805
Title: A Phase 2b, Randomized, Double-Blind, Multicenter, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Pharmacokinetics of Treprostinil Palmitil Inhalation Powder in Participants With Pulmonary Arterial Hypertension
Brief Title: A Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Treprostinil Palmitil Inhalation Powder in Participants With Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insmed Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INS1009-202; 2021-001528-16 (EudraCT Number); 2023-505541-99-00 (Other: EU CT Number)
Record Dates: First submitted 2021-11-24; First posted 2021-12-07 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Treprostinil Palmitil; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treprostinil Palmitil Inhalation Powder (Experimental): Participants will be administered TPIP once per day at a starting dose of 80 micrograms (μg). Participants will be up-titrated to the highest tolerated dose for each individual participant of between 80 μg and 640 μg during the initial 3 weeks of treatment. The overall treatment period will be 16 weeks.
  Interventions: Drug: Treprostinil Palmitil
- Placebo (Placebo Comparator): Participants will be administered a placebo matching TPIP once per day for 16 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Treprostinil Palmitil — Administered by oral inhalation using a Plastiape capsule-based dry powder inhaler.
  Other Names: INS1009
  Arms: Treprostinil Palmitil Inhalation Powder
Drug: Placebo — Administered by oral inhalation using a Plastiape capsule-based dry powder inhaler.
  Arms: Placebo

SUMMARY:
The main objective of the study is to assess the effect of treprostinil palmitil inhalation powder (TPIP) compared with placebo on pulmonary vascular resistance.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be ≥ 18 to ≤ 75 years at the time of signing the informed consent form (ICF).
* Participants must have a diagnosis of World Health Organization (WHO) Group 1 Pulmonary Hypertension (PH) [pulmonary arterial hypertension (PAH)] in any of the following subtypes:

  1. Idiopathic
  2. Heritable
  3. Drug/toxin-induced or connective tissue disease (CTD)-associated PAH
  4. Congenital heart disease-related with simple systemic-to-pulmonary shunt at least 1 year following repair.
* PAH diagnosis for at least 3 months.
* Participants must be on stable PH therapy consisting of up to 2 medications from the following classes:

  1. Endothelin receptor antagonists (eg, ambrisentan, bosentan, macitentan)
  2. Phosphoesterase type 5 inhibitors (eg, sildenafil, tadalafil)
  3. Guanylate cyclase stimulator (eg, riociguat)
* No change in PH medications (eg, ambrisentan, bosentan, macitentan, sildenafil, tadalafil, riociguat) or dosage for at least 30 days prior to Screening.
* No change in long-term diuretic use or dosage for at least 30 days prior to Screening.
* Body Mass Index (BMI) within the range 18.0-37.0 kg/m^2 (inclusive).
* Male participants: Male participants who are not sterile and have female partners of childbearing potential, must be using effective contraception from Day 1 to at least 90 days after the last dose of study drug.
* Female participants: Women must be postmenopausal (defined as no menses for 12 months without an alternative medical cause), surgically sterile, (ie, post-tubal ligation for at least 12 months) or using highly effective contraception methods (ie, methods that alone or in combination achieve <1% unintended pregnancy rates per year when used consistently and correctly) from Day 1 to at least 90 days after the last dose of study drug.
* Male participants with pregnant or non-pregnant woman of childbearing potential partner must use a condom in order to avoid potential exposure to embryo/fetus.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the ICF and in the protocol.

Exclusion Criteria:

* History of PH other than idiopathic, hereditary, drug/toxin-induced, repaired simple congenital heart disease, or CTD-associated PAH (eg, complex, congenital heart disease-associated PAH, portal hypertension-associated PAH, PH belonging to Groups 2 through 5).
* Allergy, or documented hypersensitivity or contraindication, to TPIP or Treprostinil or mannitol (an excipient of the TPIP formulation).
* Any known ventricular or supraventricular tachyarrhythmia except for paroxysmal atrial fibrillation and any symptomatic bradycardia.
* History of heart disease including left ventricular ejection fraction (LVEF) ≤ 40% or clinically significant valvular, constrictive, or symptomatic atherosclerotic heart disease (eg, stable angina, myocardial infarction, etc).
* Participation in a cardio-pulmonary rehabilitation program within 1 month of Screening Visit.
* Evidence of thromboembolic disease as assessed by ventilation-perfusion (VQ) scan, pulmonary angiography, or pulmonary computed tomography (CT) scan.
* Active liver disease or hepatic dysfunction.
* History of HIV infection.
* Established diagnosis of hepatitis B viral infection, or positive for hepatitis B surface antigen (HBsAg) at the time of Screening.
* Established diagnosis of hepatitis C viral infection at the time of screening.
* Active and current symptomatic coronavirus disease 2019 (COVID-19) or previous severe disease and/or hospitalization due to COVID-19.
* Use of live attenuated vaccines within 30 days of the Screening Visit.
* Participants with Down's Syndrome.
* History of abnormal bleeding or bruising.
* History of solid organ transplantation.
* Known or suspected immunodeficiency disorder, including history of invasive opportunistic infections (eg, tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis) despite infection resolution, or otherwise recurrent infections of abnormal frequency, or prolonged infections suggesting an immune compromised status, as judged by the Investigator.
* History of alcohol or drug abuse within 6 months prior to Screening.
* Acute or chronic impairment (other than dyspnea), limiting the ability to comply with study requirements, in particular with 6-minute walk test (eg, angina pectoris, claudication, musculoskeletal disorder, need for walking aids).
* Participants with current or recent (past 30 days) lower respiratory tract infection.
* History of malignancy in the past 5 years, with exception of completely treated in situ carcinoma of the cervix and completely treated non-metastatic squamous or basal cell carcinoma of the skin.
* Change in PH medication (endothelin receptor agonists, phosphoesterase type 5 inhibitors, and guanylate cyclase stimulators or diuretics) between Screening and Baseline.
* Have participated in any other interventional clinical studies within 30 days prior to Screening.
* Current use of cigarettes (as defined by Centers for Disease Control and Prevention) or e-cigarettes.
* Participants who currently inhale marijuana (recreational or medical).
* Pregnant or breastfeeding.

Note: Other inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2025-03-27 (Actual); Study Completion 2025-03-27 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Pulmonary Vascular Resistance at Week 16 | Baseline to Week 16

SECONDARY OUTCOMES:
Change from Baseline in 6-Minute Walk Test Distance at Week 5, Week 10 and Week 16 | Baseline and Week 5, Week 10 and Week 16
Percent Change from Baseline in 6-Minute Walk Test Distance at Week 5, Week 10 and Week 16 | Baseline and Week 5, Week 10 and Week 16
Number of Participants Who Experience a Treatment-emergent Adverse Event (AE) | Day 1 up to Week 20
Number of Participants Who Experience a Clinically Significant Change from Baseline in Clinical Laboratory Evaluations | Baseline to Week 16
Number of Participants Who Experience a Clinically Significant Change from Baseline in Vital Sign Measurements | Baseline to Week 16
Number of Participants Who Experience a Clinically Significant Change from Baseline in Electrocardiogram (ECG) Measurements | Baseline to Week 16
Number of Participants Who Experience a Clinically Significant Change from Baseline in Physical Examinations | Baseline to Week 16
Maximum Plasma Concentration (Cmax) of Treprostinil Palmitil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Maximum Plasma Concentration (Cmax) of Treprostinil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Time to Maximum Plasma Concentration (Tmax) of Treprostinil Palmitil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Time to Maximum Plasma Concentration (Tmax) of Treprostinil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Area Under the Concentration-time Curve from Time 0 to 24 Hours Post-Dose (AUC24) of Treprostinil Palmitil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Area Under the Concentration-time Curve from Time 0 to 24 Hours Post-Dose (AUC24) of Treprostinil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Area Under the Concentration-time Curve from Time 0 to Infinity (AUC∞) of Treprostinil Palmitil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Area Under the Concentration-time Curve from Time 0 to Infinity (AUC∞) of Treprostinil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Area Under the Concentration-time Curve from Time 0 to Last Measurable Concentration (AUClast) of Treprostinil Palmitil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Area Under the Concentration-time Curve from Time 0 to Last Measurable Concentration (AUClast) of Treprostinil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Apparent Total Clearance (CL/F) of Treprostinil Palmitil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Apparent Total Clearance (CL/F) of Treprostinil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Apparent Volume of Distribution After Non-Intravenous Administration (Vd/F) of Treprostinil Palmitil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Apparent Volume of Distribution After Non-Intravenous Administration (Vd/F) of Treprostinil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Elimination Half-Life (t1/2) of Treprostinil Palmitil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Elimination Half-Life (t1/2) of Treprostinil | Day 1, Weeks 2, 3, 5, 10, and 16: Predose and 0.5, 1, 2 ,4 and 6 hours post-dose
Change from Baseline in the Concentration of N-Terminal-Pro Hormone Brain Natriuretic Peptide (NT-proBNP) Levels at Week 5, Week 10 and Week 16 | Baseline and Week 5, Week 10 and Week 16 or end of study

CONTACTS AND LOCATIONS:
Locations (92):
- United States (21):
  - USA025, Phoenix, Arizona
  - USA022, Scottsdale, Arizona
  - USA021, Tucson, Arizona
  - USA023, Sacramento, California
  - USA002, West Hollywood, California
  - USA008, Gainesville, Florida
  - USA005, Jacksonville, Florida
  - USA007, Orlando, Florida
  - USA011, Tampa, Florida
  - USA010, Winter Park, Florida
  - USA009, Atlanta, Georgia
  - USA006, Chicago, Illinois
  - USA001, Chicago, Illinois
  - USA013, Indianapolis, Indiana
  - USA014, Iowa City, Iowa
  - USA003, Kansas City, Kansas
  - USA102, New York, New York
  - USA017, New York, New York
  - USA016, Dallas, Texas
  - USA012, Denison, Texas
  - USA018, Houston, Texas
- Argentina (7):
  - ARG009, Quilmes, Buenos Aires
  - ARG002, Rosario, Santa Fe Province
  - ARG006, Rosario, Santa Fe Province
  - ARG007, San Miguel de Tucumán, Tucumán Province
  - ARG004, Córdoba
  - ARG001, Córdoba
  - ARG008, Cuiudad Autónoma de Buenos Aires
- Australia (5):
  - AUS005, New Lambton Heights, New South Wales
  - AUS004, Milton, Queensland
  - AUS001, Woolloongabba, Queensland
  - AUS003, Adelaide, South Australia
  - AUS002, Hobart, Tasmania
- Austria (2):
  - AUT002, Linz, Upper Austria
  - AUT001, Vienna
- Belgium (3):
  - BEL003, Anderlecht, Brussels Capital
  - BEL002, Leuven, Vlaams Brabant
  - BEL001, Liège
- Brazil (6):
  - BRA003, Belo Horizonte, Minas Gerais
  - BRA004, Belo Horizonte, Minas Gerais
  - BRA007, Passo Fundo, Rio Grande do Sul
  - BRA006, Porto Alegre, Rio Grande do Sul
  - BRA002, Blumenau, Santa Catarina
  - BRA001, São Paulo
- DNK001, Aarhus N, Central Jutland, Denmark
- Germany (6):
  - GER005, Heidelberg, Baden-Wurttemberg
  - GER006, Dresden, Saxony
  - GER001, Halle, Saxony-Anhalt
  - GER002, Lübeck, Schleswig-Holstein
  - GER007, Berlin
  - GER003, Munich
- Italy (6):
  - ITA003, Napoli, Campania
  - ITA006, Milan, Lombardy
  - ITA005, Monza, Lombardy
  - ITA002, Pavia, Lombardy
  - ITA001, Palermo, Sicily
  - ITA004, Roma
- Japan (9):
  - JPN005, Sapporo, Hokkaidô
  - JPN004, Sapporo, Hokkaidô
  - JPN007, Kurume-Shi, Hukuoka
  - JPN006, Tsukuba, Ibaraki
  - JPN001, Kagoshima, Kagoshima-ken
  - JPN009, Nagasaki, Nagasaki
  - JPN002, Okayama, Okayama-ken
  - JPN008, Shinjuku-Ku, Tokyo
  - JPN003, Suita-Shi, Ôsaka
- Malaysia (4):
  - MYS005, Alor Star, Kedah
  - MYS002, Kuantan, Pahang
  - MYS003, Kajang, Selangor
  - MYS004, Sungai Buloh, Selangor
- Mexico (4):
  - MEX005, Lomas de Guevara, Jalisco
  - MEX003, Mexico City, Mexico City
  - MEX004, San Luis Potosí City
  - MEX001, Sertoma
- Philippines (2):
  - PHL001, Quezon City, National Capital Region
  - PHL002, Makati City
- Serbia (3):
  - SRB004, Belgrade, Belgrade
  - SRB001, Belgrade
  - SRB003, Belgrade
- Spain (7):
  - ESP006, Palma de Mallorca, Balearic Islands
  - ESP001, Santander, Cantabria
  - ESP002, Barcelona
  - ESP007, Las Palmas
  - ESP008, Madrid
  - ESP003, Seville
  - ESP004, Toledo
- CHE002, Lausanne, Vaud (fr), Switzerland
- United Kingdom (5):
  - GBR001, Bath, Avon
  - GBR002, Glasgow, Lanarkshire
  - GBR006, London, London, City of
  - GBR003, Newcastle upon Tyne, Tyne and Wear
  - GBR004, London

IPD SHARING:
Plan to Share IPD: No